CLINICAL TRIAL: NCT03807596
Title: Adjunctive Use Of Hyaluronic Acid With Scaling & Root Planing In Treatment of Chronic Periodontitis Patients With Diabetes Mellitus Type 2: A Randomized Controlled Trial
Brief Title: Hyaluronic Acid With Scaling & Root Planing In Chronic Periodontitis Patients With Diabetes Mellitus Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gihane Gharib Madkour, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15062011
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP group (Active Comparator): Chronic periodontitis patients with type 2 diabetes mellitus recieved Periodontal treatment in the form of scaling & root planing (SRP) alone.
  Interventions: Procedure: Scaling & root planning alone
- Hyaluronic acid & SRP group (Experimental): Chronic periodontitis & type 2 diabetes mellitus patients received Periodontal treatment in the form of scaling & root planing (SRP) with the adjunctive use of hyaluronic acid.
  Interventions: Procedure: Periodontal treatment with Hyaluronic acid associated with SRP

INTERVENTIONS:
Procedure: Periodontal treatment with Hyaluronic acid associated with SRP — In addition to SRP, patients in the test group received adjunct subgingival application of hyaluronic acid in all selected periodontal pockets.
  Arms: Hyaluronic acid & SRP group
Procedure: Scaling & root planning alone — Patients received full-mouth supra- & sub-gingival SRP with the use of ultrasonic device & periodontal universal & Gracey curettes under local anesthesia.
  Arms: SRP group

SUMMARY:
The present study aimed to assess the adjunctive use of Hyaluronic acid with scaling & root planing (SRP) in patients with chronic periodontitis & diabetes mellitus type 2.

DETAILED DESCRIPTION:
Thirty subjects with chronic periodontitis & diabetes mellitus type 2 were included in this randomized clinical trial. These subjects were randomly allocated into test & control equal groups. The test group comprised fifteen patients who received SRP with subgingival application of Hyaluronic acid as an adjunct. The control group included fifteen patients who received SRP alone. Plaque index (PI), gingival index (GI), probing depth (PD) & clinical attachment level (CAL) were measured & documented at baseline, 6 weeks & 12 weeks intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic periodontitis and type 2 diabetes mellitus
* Minimum of 20 teeth
* Clinical attachment level (CAL) ≥ 3 mm
* Probing depth (PD) ≥ 4 mm.

Exclusion Criteria:

* Pregnant females
* Smokers

Ages: 38 Months to 56 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Gain in clinical attachment level | 12 weeks
  Gain in clinical attachment level will be measured in millimeter by William's graduated periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Gihane G Madkour, Ass Prof, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No